CLINICAL TRIAL: NCT03364231
Title: A Phase 2 Study to Assess the Efficacy and Safety of TGR-1202 (Umbralisib) Monotherapy in Patients With Non-Follicular Indolent Non-Hodgkin's Lymphoma
Brief Title: Study to Assess the Efficacy and Safety of Umbralisib in Participants With Non-Follicular Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-1202-202
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia; Non Follicular Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Marginal Zone Lymphoma (MZL): Umbralisib (Experimental): Participants with non-follicular indolent non-Hodgkin's lymphoma (iNHL) with MZL as the histology type received umbralisib, 800 milligrams (mg), orally, once daily (QD), until disease progression, unacceptable toxicity, or withdrawal from the study whichever occurred first.
  Interventions: Drug: Umbralisib
- Waldenstrom's Macroglobulinemia (WM): Umbralisib (Experimental): Participants with non-follicular iNHL with WM as the histology type received umbralisib, 800 mg, orally, QD, until disease progression, unacceptable toxicity, or withdrawal from the study whichever occurred first.
  Interventions: Drug: Umbralisib

INTERVENTIONS:
Drug: Umbralisib — Oral Daily Dose
  Other Names: TGR-1202

SUMMARY:
This research study will evaluate the safety and efficacy of a study drug called Umbralisib (also known as TGR-1202) alone as a possible treatment for Waldenstrom's Macroglobulinemia that has come back or that has not responded to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Waldenstroms Macroglobulinemia
* Relapsed or refractory after at least one prior treatment regimen
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Evidence of hepatitis B virus, hepatitis C virus or known HIV infection
* Prior autologous stem cell transplant within 6 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cheson, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (4):
- United States (4):
  - TG Therapeutics Investigational Trial Site, Washington D.C., District of Columbia
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 21 participants were enrolled at 4 investigative centers across the United States from 30 November 2017 to 15 February 2022.
Groups:
- Marginal Zone Lymphoma (MZL): Umbralisib: Participants with non-follicular indolent non-Hodgkin's lymphoma (iNHL) with MZL as the histology type received umbralisib, 800 milligrams (mg), orally, once daily (QD), until disease progression, unacceptable toxicity or withdrawal from the study whichever occurred first.
Period: Overall Study
Arm/Group | Marginal Zone Lymphoma (MZL): Umbralisib | Waldenstrom's Macroglobulinemia (WM): Umbralisib
Started | 8 | 13
Safety Population (Safety population included all enrolled participants who received at least one dose of study treatment.) | 8 | 13
Modified Intent-To-Treat (mITT) (mITT population included all participants who received at least one dose of study treatment and provided at least some post baseline efficacy assessment.) | 8 | 10
Completed | 0 | 0
Not Completed | 8 | 13
Not completed — Adverse Event | 1 | 4
Not completed — Death | 1 | 0
Not completed — Investigator Decision | 2 | 2
Not completed — Sponsor Discontinuation of the Study | 2 | 1
Not completed — Withdrawal of Subject Consent | 1 | 0
Not completed — Reason Not Specified | 1 | 0
Not completed — Disease Progression | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of study treatment.
Groups:
- MZL: Umbralisib: Participants with non-follicular iNHL with MZL as the histology type received umbralisib, 800 mg, orally, QD, until disease progression, unacceptable toxicity, or withdrawal from the study whichever occurred first.
- WM: Umbralisib: Participants with non-follicular iNHL with WM as the histology type received umbralisib, 800 mg, orally, QD, until disease progression, unacceptable toxicity, or withdrawal from the study whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | MZL: Umbralisib | WM: Umbralisib | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.64) | 67.7 (5.78) | 69.3 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 11 | 17
  Black or African American | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed by Revised Response Criteria for Non- Hodgkin's Lymphoma (Lugano Classification) and Consensus-Based 6th International Workshop on Waldenstrom's Macroglobulinemia (IWWM)
Description: ORR for MZL=percentage of participants with complete response (CR)/partial response (PR). ORR for WM=CR/PR/very good partial response (VGPR)/minor response (MR). Response assessed per revised Lugano Classification for MZL &per IWWM for WM participants. Per Lugano criteria CR=complete disappearance of all evidence of disease & disease-related symptoms. PR=regression of measurable disease & no new disease sites. Regression=≥50% decrease in the sum of the products of the diameters (SPD) of index lesions, with no increase in size of other lymph nodes/liver/spleen.Per IWWM criteria CR=disappearance of serum monoclonal immunoglobulin M (IgM) protein by immunofixation with a normal serum IgM level. VGPR=reduction of monoclonal IgM protein >90% from baseline. PR=reduction of monoclonal IgM protein between 50-90% from baseline with regression of measurable disease. Regression defined in similar manner as Lugano Classification. MR=reduction of monoclonal IgM protein >25% but <50% from baseline.
Time Frame: Every 3 cycles (1 Cycle = 28 days) from Day 1 Cycle 1 up to approximately 4.2 years
Population: mITT population included all participants who received at least one dose of study treatment and provided at least some post baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 8 | 10
percentage of participants | 37.5 [8.5 to 75.5] | 30.0 [6.7 to 65.2]

2. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from documentation of a response to treatment to the first documentation of tumor progression or death due to any cause, whichever comes first.
Time Frame: From the first demonstration of response to umbralisib till disease progression/death (up to approximately 4.2 years)
Population: mITT population included all participants who received at least one dose of study treatment and provided at least some post baseline efficacy assessment. 'Overall number of participants analyzed' is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: months
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 3 | 3
months | 21.2 [3 to 33] | 13 [5 to 14]

3. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate is defined as percentage of participants who achieved CR. CR was assessed using Revised Response Criteria for Non- Hodgkin's Lymphoma (Lugano Classification) for participants with MZL and Consensus-Based 6th IWWM for participants with WM.
  Per Lugano Classification, CR= the complete disappearance of all evidence of disease and disease-related symptoms i.e., liver/spleen non palpable and normal in size and disappearance of nodules related to lymphoma.
  Per IWWM criteria, CR=disappearance of serum monoclonal IgM protein by immunofixation with a normal serum IgM level, liver/spleen non palpable and normal in size and disappearance of nodes related to WM.
Time Frame: Every 3 cycles (1 Cycle = 28 days) from Day 1 Cycle 1 up to approximately 4.2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 8 | 10
percentage of participants | 12.5 [0.3 to 52.7] | 0 [NA to NA] — Since none of the participants had a complete response, 95% CI could not be calculated.

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the interval from Cycle 1 (1 cycle = 28 days) Day 1 to the earlier of the first documentation of definitive disease progression or death from any cause. Assessment of progressive disease (PD) was based on Revised Response Criteria for non-Hodgkin's lymphoma, Lugano Classification for participants with MZL and consensus-based 6th IWWM for participants with WM.
  Per Lugano Classification, PD was defined as the appearance of any new lesion more than 1.5 centimeters (cm) in any axis, even if other lesions are decreasing in size. At least a 50% increase from nadir in one of the following: SPD of index lesions, greatest transverse diameter (GTD) of any individual previously involved node, or GTD of any previously involved node provided that the GTD of that node is now ≥ 1.5 cm.
  Per IWWM criteria participants, PD was defined as more than 25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable to the disease.
Time Frame: From date of randomization until the date of first documented progression (up to approximately 4.2 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 8 | 10
months | 47.1 [1.4 to 47.1] | 18.4 [2.1 to 35.0]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as a composite endpoint measuring time from Cycle 1/Day 1 to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death. PD was assessed based on Revised Response Criteria for non-Hodgkin's lymphoma, Lugano Classification for participants with MZL and consensus-based 6th IWWM for participants with WM.
  Per Lugano Classification, PD was defined as the appearance of any new lesion more than 1.5 cm in any axis, even if other lesions are decreasing in size. At least a 50% increase from nadir in one of the following: SPD of index lesions, GTD of any individual previously involved node, or GTD of any previously involved node provided that the GTD of that node is now ≥ 1.5 cm.
  Per IWWM criteria PD was defined as more than 25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable to the disease.
Time Frame: From first dose on Day 1 of Cycle 1 (28 days = 1 cycle) up to discontinuation of treatment (up to approximately 4.2 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 8 | 10
months | 13.1 [1.4 to NA] — Upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 6.5 [2.1 to 15.9]

6. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant that does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From first dose of study treatment up to end of study (up to approximately 4.2 years)
Population: Safety population included all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- MZL: Umbralisib: Participants with non-follicular iNHL with MZL as the histology type received umbralisib, 800 mg, orally, QD, until disease progression, unacceptable toxicity or withdrawal from the study whichever occurred first.
Arm/Group | MZL: Umbralisib | WM: Umbralisib
Number analyzed (Participants) | 8 | 13
Participants | 8 | 13

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to end of study (up to approximately 4.2 years)
Description: Safety population included all enrolled participants who received at least one dose of study treatment.
Arm/Group | MZL: Umbralisib | WM: Umbralisib
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/13
Other Adverse Events (participants affected / at risk) | 8/8 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MZL: Umbralisib (N=8) | WM: Umbralisib (N=13)
Colitis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MZL: Umbralisib (N=8) | WM: Umbralisib (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Nausea (Gastrointestinal disorders) | 4 | 7
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 2 | 3
Pyrexia (General disorders) | 1 | 2
Asthenia (General disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 2
Early satiety (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Mucosal disorder (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Reaction to previous exposure to any vaccine (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Decreased apetite (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspneoa (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Annular elastolytic giant cell granuloma (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Schnitzler's syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Pallor (Vascular disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03364231/Prot_SAP_000.pdf